CLINICAL TRIAL: NCT02127333
Title: Role of Acute and Chronic Hypoxemia for Vascular Function
Brief Title: Role of Oxygen for Vascular Dysfunction
Status: Completed | Type: Observational
Sponsor: Klinik für Kardiologie, Pneumologie und Angiologie (Other)
Responsible Party: Sponsor-Investigator, Klinik für Kardiologie, Pneumologie und Angiologie, Division of Cardiology, Pulmonary Diseases, Vascular Medicine, Heinrich-Heine University, Duesseldorf
Organization: Heinrich-Heine University, Duesseldorf (Other)
Other Study IDs: COPD_pO2
Record Dates: First submitted 2014-04-29; First posted 2014-04-30 (Estimated); Last update posted 2014-12-16 (Estimated); Status verified 2014-12

CONDITIONS: Endothelial Dysfunction; FMD; IMT; Microcirculation; Oxygen Pressure; Carbon Dioxide Pressure; Oxygen Saturation; Forced Expiratory Volume After 1 Second
Keywords: chronic obstructive pulmonary disease; Coronary artery disease; Endothelial function
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- CAD patients with COPD
- CAD patients without COPD
- healthy volunteers

SUMMARY:
Hypoxemia may contribute increased morbidity and mortality in chronic obstructive pulmonary disease (COPD) patients. We aim to characterize the role of acute and chronic hypoxemia for vascular function. For this purpose we measure capillary oxygen concentration and vascular.

Vascular function is assessed by flow-mediated dilation oft he brachial artery, forearm blood flow and laser doppler perfusion imaging.

We hypothesize that hypoxemia leads to impaired vascular function.

ELIGIBILITY:
Inclusion Criteria:

* stable coronary artery disease
* stable chronic obstructive pulmonary disease

Exclusion Criteria:

* acute myocardial infarction within 30 days
* acute exacerbated COPD within 30 days
* acute infections
* severe acute or chronic renal failure
* severe heart failure
* atrial fibrillation
* severe cardiac arrhythmia
* hypotension
* active malignant disease
* active rheumatic disease
* pulmonary hypertension with vasoactive therapy

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: CAD patients with or without COPD; healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2011-01; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Flow-mediated dilation of the brachial artery | Baseline

SECONDARY OUTCOMES:
Forearm blood flow | Baseline
Laser doppler perfusion | Baseline
Intima-media thickness of the brachial artery | Baseline
Fractional diameter change of the brachial artery | Baseline
Endothelium-independent vasodilation of the brachial artery | Baseline

OTHER OUTCOMES:
Plasma nitrite concentration | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Christian Heiss, MD, Principal Investigator — Division of Cardiology, Pulmonary Disease and Vascular Medicine; Malte Kelm, MD, Study Chair — Division of Cardiology, Pulmonary Disease and Vascular Medicineine
Locations (1):
- Division of Cardiology, Pulmonary Disease and Vascular Medicine, Düsseldorf, Germany

REFERENCES:
- See also: Related Info — http://www.uniklinik-duesseldorf.de/kardiologie